CLINICAL TRIAL: NCT00913640
Title: Prospective Memory in Parkinson's Disease
Acronym: ProMem
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 05-0203
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Memory; Prospective Memory; Parkinson's Disease
Keywords: Prospective Memory Performance; Prospective Memory Outcome; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PD Group
- Control Group

SUMMARY:
The investigators tested whether prospective memory is impaired in individuals with Parkinson's Disease compared to controls using reliable and validated experimental measures. Also, the investigators assessed the impact of Parkinson's medication on prospective memory performance in PD to better estimate prospective memory function in PD patients' everyday (chronically treated) life.

ELIGIBILITY:
Inclusion Criteria:

* PD Group:

  * Clinically definite PD
  * 40-70 years old
  * Hoehn and Yahr stage I,II,III
  * Currently treated with Levodopa/carbidopa
* Control Group:

  * 40-70 years old
  * Spouses of PD Group preferred

Exclusion Criteria:

* PD Group and Control Group:

  * Significant neurological problems
  * Significant current psychiatric diagnoses
  * Mini Mental Status Exam score < 24 (MMSE)
  * Any significant abnormality on brain imaging
  * MPTP exposure
  * Control Participants met the same exclusion criteria described above as well as a biological family history of PD

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Movement Disorder Clinic at Washington University St. Louis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2010-08-27 (Actual); Study Completion 2010-08-27 (Actual)

PRIMARY OUTCOMES:
Virtual Week | One session at baseline.
  Prospective Memory Task; Score range is 0-100%, with higher scores being better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Foster ER, Rose NS, McDaniel MA, Rendell PG. Prospective memory in Parkinson disease during a virtual week: effects of both prospective and retrospective demands. Neuropsychology. 2013 Mar;27(2):170-81. doi: 10.1037/a0031946. PMID 23527645